CLINICAL TRIAL: NCT03806270
Title: Hydroxyzine Dihydrochloride Premedication is a Necessity for Pediatric Patients Undergoing Strabismus Surgery; An Observational Clinical Trial Controlled With Midazolam
Brief Title: Hydroxyzine Dihydrochloride Premedication is a Necessity for Strabismus Surgery
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Fatma Ferda Kartufan, Assistant Professor, Yeditepe University
Other Study IDs: KAEK884
Record Dates: First submitted 2018-12-24; First posted 2019-01-16 (Actual); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Strabismus; Reflex, Oculocardiac; Hydroxyzine; Bradycardia Sinus
Keywords: Strabismus surgery; Oculocardiac reflex; Hydroxyzine dihydrochloride; Midazolam; Premedication; The Ramsay Scale
MeSH Terms: conditions — Strabismus | interventions — Midazolam; Hydroxyzine; Validol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Midazolam: Demizolam, once on the operation day, usually ordered 15 minutes before strabismus operation by another anesthesiologist who is charged to perform anesthesia who is not related with the trial.The maximum dose of 0.5 mg/kg midazolam is given orally with cherry juice of maximum 5 ml. in Yeditepe University Hospital to the pediatric patients by the anesthesiologists.
  In all groups patients are not selected to the groups and premedication and doses are not given by the investigator, they grouped according to the premedication given by the anesthesiologists, after the operation retrospectively.
  Interventions: Drug: Midazolam
- Midazolam&Hydroxyzine dihydrochloride1/2: Midazolam and Hydroxyzine dihydrochloride, once on the operation day, usually ordered 15 minutes before strabismus operation by another anesthesiologist who is charged to perform anesthesia who is not related with the trial.The maximum dose of 0.5 mg/kg midazolam is given orally with hydroxyzine dihydrochloride (dose of 0.5 mg/kg) in Yeditepe University Hospital to the pediatric patients by the anesthesiologists.
  In all groups patients are not selected to the groups and premedication doses are not given by the investigator, they grouped according to the premedication given by the anesthesiologists, after the operation retrospectively.
  Interventions: Drug: Midazolam; Drug: Hydroxyzine Dihydrochloride
- Midazolam&Hydroxyzine dihydrochloride: Midazolam and Hydroxyzine dihydrochloride, once on the operation day, usually ordered 15 minutes before strabismus operation by another anesthesiologist who is charged to perform anesthesia who is not related with the trial.The maximum dose of 0.5 mg/kg midazolam is given orally with the maximum dose of 1mg/kg hydroxyzine dihydrochloride in Yeditepe University Hospital to the pediatric patients by the anesthesiologists.
  In all groups patients are not selected to the groups and premedication doses are not given by the investigator, they grouped according to the premedication given by the anesthesiologists, after the operation retrospectively.
  Interventions: Drug: Midazolam; Drug: Hydroxyzine Dihydrochloride

INTERVENTIONS:
Drug: Midazolam — Demizolam 15mg/ml ampules, given orally with cherry juice
  Other Names: Dormicum,8699505751689,N05CD08; Demizolam,8699769750077,N05CD08; Zolamide,8680184750025,N05CD08
Drug: Hydroxyzine Dihydrochloride — Atarax 2mg/ml syrup, given orally
  Other Names: ATARAX 200 ml syrup,8699624570062,N05BB01; VALIDOL,8699705590019,N05BB01
  Groups: Midazolam&Hydroxyzine dihydrochloride; Midazolam&Hydroxyzine dihydrochloride1/2

SUMMARY:
Oculocardiac reflex (OCR) is usually happening in pediatric strabismus surgery and observed just when the surgent pulls the ocular muscles. The reflex is one of the trigemino-vagal reflexes, and causes bradycardia, arrhythmia, and even cardiac arrest during eye surgery.

Premedication for relaxation with drugs like hydroxyzine dihydrochloride or midazolam before surgery of the pediatric population is often used in Turkey, although it is not recommended in foreign countries. Some recent studies showed that when midazolam and hydroxyzine dihydrochloride used together not only, they lessen agitation before surgery but also they prevent emergence agitation.

The primary aim of this prospective observational study is to show the effect of hydroxyzine dihydrochloride on preventing the pediatric patient from Oculocardiac reflex related to strabismus surgery.

DETAILED DESCRIPTION:
Strabismus surgery is a frequently performed surgery in the Turkish population from one year of age to adults. Oculocardiac reflex(OCR) is the most recent complication happens during the operation, and it occurs approximately 20% to 80% according to its definition, in strabismus surgery.

OCR is defined as the presence of dysrhythmia or a sudden heart rate decreased by 20% after traction on the extraocular muscles. OCR is one of the trigemino-vagal reflexes and causes bradycardia, arrhythmia and even cardiac arrest during eye surgery. To prevent patients from this complication the operator and anesthesiologist must cooperate during the operation because the first treatment is to stop traction of the muscle, the second one is to use atropine after diagnosing bradycardia.

Oculocardiac reflex related trials were done for decades; searching for how and when it happens, which ocular muscles are related mostly, or which patients are at risk of OCR( age, heart rate related) are the most researched ones. According to our knowledge, there is no research about a premedication to prevent OCR during strabismus surgery.

Before this study has planned by the investigator, the investigator had seen many OCR occurrence related to strabismus surgery, treated either with pausing the surgery or with atropin intravenous utilization in other clinics. After started working in this university hospital the investigator recognized those pediatric patients whom premedicated do not need to treat in the strabismus surgery because the OCR incidence was decreased dramatically. The investigator has planned this observational research at Yeditepe University Hospital because in this hospital pediatric patients receive variable oral premedication for sedation before surgery and for the prevention of emerging agitation. In Yeditepe University Hospital oral premedication( with variable drugs and variable doses) is nearly always ordered by anesthesiologists unless there is a comorbidity or allergy anamnesis related to the drugs planning to use.

This current study is planned as observational. The investigator does not allow to give any orders about premedications or treatments before or during strabismus surgery. The Induction and the maintenance of anesthesia are also variable because there is no intervening to the anesthetist who performs anesthesia. The anesthetist who orders the premedication and performs anesthesia during strabismus surgery is not related to the trial and do not know the aim of the trial.

The investigator is informed about the surgery on the day of the operation. The investigator and the patient's encounter before the study are about having the written consent form after explanation of the study. The only time to discriminate the patient from the study, by the anamnesis of the patient that is taken (about any comorbidities) during the encounter, according to the trials eligibility criteria if the patient and the patient has approved for including the trial. The investigator has even no permission to access the demographic data of the patient from the clinical papers which nurses have prepared because the investigator is not the anesthesiologist of the patient. Therefore the demographic data of the patient and the premedication performed to the patient is recorded after the operation retrospectively as the ethical committee approved. So, this current trial is not randomized, and there is no placebo group also, as a control group which is needed for an interventional one. Patients included to this trial were grouped after the end of the operation according to the premedication utilized, while the patient is awake in the service room after the operation, by having permission to access the demographic data and the premedication that had utilized before operation retrospectively.

The prospective part of this study is planned to perform in the operation theatre observationally without knowing which premedication is utilized to the patient. In the operation theatre, the investigator observes the patient coming to the operation theatre and records the patients Ramsey Sedation Score before the operation starts. The heart rate 1, the heart rate 2 and the heart rate 3 data are planned to be recorded from the EKG monitorisation of the patient; in cooperation with the operator( the operator warns the investigator before the traction of the orbital muscle and informs about the name of the orbital muscle.). The investigator calculates the difference between the heart rate3 and heart rate2 and records if OCR occurred or not. If OCR occurred, the investigator observes and records how it is treated by the anesthesiologist in the operation theatre and the orbital muscle name which OCR occurred during its traction. The investigator is also not allowed to order any treatment about OCR during the operation. Because it is hard to plan this kind of an observational study the investigator had two years of paperwork to explain the planning of this observational study to be approved from both "Yeditepe University Clinical Trials Ethical Committee," and from "The Turkish Ministry of health, Turkish Medicines and Medical Devices Agency." A medical doctor from another clinic is charged with the monitorisation of this clinical trial by the ethical committee of the Yeditepe University whose identity is not known by the investigator.

The primary aim of this prospective observational trial is to compare three different premedication methods observationally, to see if there is any difference in the OCR occurrence in strabismus surgery. The secondary aim is to compare the Ramsey Sedation Scores of the patients before surgery, the heart rates during the operation and their effect on OCR.

The hypothesis is that; the pediatric patients premedicated with hydroxyzine dihydrochloride would be prevented from OCR during strabismus surgery because of the drug's side-effect of tachycardia while they are sedated before surgery as a positive effect.

ELIGIBILITY:
Inclusion Criteria:

* Strabismus, surgery needed
* Esotropia, surgery needed

Exclusion Criteria:

* Chronic disease
* Arrhythmia
* Glaucoma(narrow-angle)

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged between 1 to 10 years who are diagnosed as strabismus or esotropia, and scheduled for strabismus surgery.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ferda F Kartufan, Assist.Prof, Principal Investigator — Yeditepe University Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Yeditepe University Ophtalmology Research Center, Istanbul, Beşiktaş
  - Yeditepe University Hospital, Istanbul, İçerenköy

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared.

REFERENCES:
- [Background] Oh JN, Lee SY, Lee JH, Choi SR, Chin YJ. Effect of ketamine and midazolam on oculocardiac reflex in pediatric strabismus surgery. Korean J Anesthesiol. 2013 Jun;64(6):500-4. doi: 10.4097/kjae.2013.64.6.500. Epub 2013 Jun 24. PMID 23814649
- [Background] Koner O, Ture H, Mercan A, Menda F, Sozubir S. Effects of hydroxyzine-midazolam premedication on sevoflurane-induced paediatric emergence agitation: a prospective randomised clinical trial. Eur J Anaesthesiol. 2011 Sep;28(9):640-5. doi: 10.1097/EJA.0b013e328344db1a. PMID 21822077
- [Derived] Kartufan FF, Kizilcik N, Ziylan S, Menda F. Hydroxyzine Dihydrochloride Premedication Is a Necessity for Pediatric Patients Undergoing Strabismus Surgery: An Observational Prospective Clinical Trial. J Ophthalmol. 2022 Sep 21;2022:4137144. doi: 10.1155/2022/4137144. eCollection 2022. PMID 36189149

RESULTS

PARTICIPANT FLOW:
Groups:
- Midazolam: Demizolam, once on the operation day, usually ordered 15 minutes before strabismus operation by another anesthesiologist who is charged to perform anesthesia who is not related with the trial.The maximum dose of 0.5 mg/kg midazolam is given orally with cherry juice of maximum 5 ml. in Yeditepe University Hospital to the pediatric patients by the anesthesiologists.
  In all groups patients are not selected to the groups and premedication and doses are not given by the investigator, they grouped according to the premedication given by the anesthesiologists, after the operation retrospectively.
  Midazolam: Demizolam 15mg/ml ampules, given orally with cherry juice
- Midazolam&Hydroxyzine dihydrochloride1/2: Midazolam and Hydroxyzine dihydrochloride, once on the operation day, usually ordered 15 minutes before strabismus operation by another anesthesiologist who is charged to perform anesthesia who is not related with the trial.The maximum dose of 0.5 mg/kg midazolam is given orally with hydroxyzine dihydrochloride (dose of 0.5 mg/kg) in Yeditepe University Hospital to the pediatric patients by the anesthesiologists.
  In all groups patients are not selected to the groups and premedication doses are not given by the investigator, they grouped according to the premedication given by the anesthesiologists, after the operation retrospectively.
  Midazolam: Demizolam 15mg/ml ampules, given orally with cherry juice
  Hydroxyzine Dihydrochloride: Atarax 2mg/ml syrup, given orally
- Midazolam&Hydroxyzine Dihydrochloride: Midazolam and Hydroxyzine dihydrochloride, once on the operation day, usually ordered 15 minutes before strabismus operation by another anesthesiologist who is charged to perform anesthesia who is not related with the trial.The maximum dose of 0.5 mg/kg midazolam is given orally with the maximum dose of 1mg/kg hydroxyzine dihydrochloride in Yeditepe University Hospital to the pediatric patients by the anesthesiologists.
  In all groups patients are not selected to the groups and premedication doses are not given by the investigator, they grouped according to the premedication given by the anesthesiologists, after the operation retrospectively.
  Midazolam: Demizolam 15mg/ml ampules, given orally with cherry juice
  Hydroxyzine Dihydrochloride: Atarax 2mg/ml syrup, given orally
Period: Overall Study
Arm/Group | Midazolam | Midazolam&Hydroxyzine dihydrochloride1/2 | Midazolam&Hydroxyzine Dihydrochloride
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Midazolam&Hydroxyzine dihydrochloride1/2 | Midazolam&Hydroxyzine Dihydrochloride | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 15 | 45
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.3 (2.5) | 3.5 (2.2) | 2.9 (1.8) | 4.2 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 8 | 21
  Male | 10 | 7 | 7 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 15 | 15 | 15 | 45
Region of Enrollment [Number; unit: participants]
  Turkey | 15 | 15 | 15 | 45
Heart Rate 1 [Mean (Standard Deviation); unit: beats per minute] | 114.4 (22.1) | 125.8 (13.5) | 122.33 (13.7) | 120.8 (17.2)

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate-1
Description: The lowest heart rate observed from EKG monitorization at the "time-out" after the anesthesia induction, and just before the surgery starts. Heart rate-1 is a data, not an assessing change, which is recoded during the "time-out". "The time-out" is when the patient's name, the procedure, the surgent name is repeated before the operation starts.
Time Frame: 1 minute, at the "time out", through study completion an average of 6 months
Population: Heart Rate1 was measured from each of the 45 participants, during "time-out" right after anesthesia induction and before surgery begins. This measurement is not related to orbital muscle traction.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Midazolam | Midazolam&Hydroxyzine dihydrochloride1/2 | Midazolam&Hydroxyzine Dihydrochloride
Number analyzed (Participants) | 15 | 15 | 15
beats per minute | 114.4 (22.1) | 125.8 (13.5) | 122.3 (13.7)

2. Primary Outcome: Heart Rate-2
Description: The heart rate observed from EKG monitorization at the time operator warns the investigator just before the traction of the orbital muscle. Heart rate-2 is a data, not an assessing change, which is recorded during the operation at the time operator warns. The heart rate observed from EKG monitorization, before every orbital muscle traction at the time the operator's warning before traction.
Time Frame: 1 minute, at the strabismus surgery operation, through study completion an average of 6 months
Population: "Orbital muscles" which surgery performed. It is not equal to the participant number. Related to strabismus surgery, the number of muscles surgery performed on a participant might change; like as one eye 2 muscles, two eyes but 1 muscle for each eye or two eyes 2 muscle for each.
Measure: Mean (Standard Deviation); unit: beats per minute
Units Other Than Participants: Orbital Muscles
Arm/Group | Midazolam | Midazolam&Hydroxyzine dihydrochloride1/2 | Midazolam&Hydroxyzine Dihydrochloride
Number analyzed (Participants) | 15 | 15 | 15
Number analyzed (Orbital Muscles) | 29 | 28 | 30
beats per minute | 110.4 (14.1) | 125.3 (13.1) | 124.8 (11.9)

3. Primary Outcome: Heart Rate-3
Description: The lowest heart rate observed from EKG monitorization, after every orbital muscle traction within 120 seconds. Heart rate-3 is a data, not an assessing change, which is recorded within 120 seconds after traction applied.
Time Frame: within 120 seconds after the orbital muscle traction, at the strabismus surgery operation, through study completion an average of 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute
Units Other Than Participants: Orbital Muscles
Arm/Group | Midazolam | Midazolam&Hydroxyzine dihydrochloride1/2 | Midazolam&Hydroxyzine Dihydrochloride
Number analyzed (Participants) | 15 | 15 | 15
Number analyzed (Orbital Muscles) | 29 | 28 | 30
beats per minute | 90.8 (16.6) | 113.4 (15.6) | 117.9 (12.7)

4. Primary Outcome: Number of Observed Oculocardiac Reflex(OCR)
Description: The OCR is a heartbeat anomaly(bradycardia, any arrhythmia, or cardiac arrest) associated with traction applied to the extraocular muscles during strabismus surgery. The specific criteria were as follows: the lowest heart rate observed within 120 seconds from EKG monitorization, after every orbital muscle traction, was less than 20% of the heart rate observed directly preceding traction of the orbital muscle. Additionally, any kind of arrhythmia or cardiac arrest occurrence within 120 seconds after orbital muscle traction was also defined as an OCR.
Time Frame: 2 minutes, at the strabismus surgery operation after recording Heart Rate-3, through study completion an average of 6 months
Population: OCR occurrence (0: no and 1: yes) was recorded for every orbital muscle. So it is not equal to the participant number.
Measure: Count of Units; unit: orbital muscles
Units Other Than Participants: orbital muscles
Arm/Group | Midazolam | Midazolam&Hydroxyzine dihydrochloride1/2 | Midazolam&Hydroxyzine Dihydrochloride
Number analyzed (Participants) | 15 | 15 | 15
Number analyzed (orbital muscles) | 29 | 28 | 30
orbital muscles | 15 | 6 | 1

5. Secondary Outcome: Ramsay Sedation Score
Description: If Awake; Ramsay 1: Anxious, agitated, restless; Ramsay 2: Cooperative, oriented, tranquil; Ramsay 3: Responsive to commands only If Asleep; Ramsay 4: Brisk response to a light glabellar tap or loud auditory stimulus;
  Ramsay 5: Sluggish response to a light glabellar tap or loud auditory stimulus; Ramsay 6:
  No response to a light glabellar tap or loud auditory stimulus
Time Frame: After patient transferred into the operation theatre and before anesthesia induction, through study completion an average of 6 months
Population: every participant that had only midazolam or one of the midazolam and hydroxizine premedications before surgery. Ramsay sedation score is evaluated by the investigator before surgery, in the operating theatre without knowing which premedication was utilized to the participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Midazolam&Hydroxyzine dihydrochloride1/2 | Midazolam&Hydroxyzine Dihydrochloride
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Ramsay 1 | 2 | 0 | 2
  Ramsay 2 | 13 | 15 | 9
  Ramsay 3 | 0 | 0 | 4
  Ramsay 4 | 0 | 0 | 0
  Ramsay 5 | 0 | 0 | 0
  Ramsay 6 | 0 | 0 | 0

6. Other Pre Specified Outcome: Number of Orbital Muscles of the Participants With Different Considerations Taken With Respect to the Treatment of OCR
Description: The investigator records every OCR treatment like; pausing surgery, atropin 20mcg/kg intravenous treatment or cardiac resuscitation.
Time Frame: within 5 minutes after defining the OCR occurrence, at the strabismus surgery operation, through study completion an average of 6 months
Population: midazolam group includes 15 participants; total 29 orbital muscles operated, in 15 of them OCR occurred.
  Midazolam&Hydroxyzine1/2 group includes 15 participants; total 28 orbital muscles operated, in 6 of them OCR occurred.
  Midazolam&Hydroxyzine group includes 15 participants; total 30 orbital muscles operated, in 1 of them OCR occurred.
Measure: Number; unit: number of orbital muscle/s, OCR occured
Units Other Than Participants: number of orbital muscle/s, OCR occured
Arm/Group | Midazolam | Midazolam&Hydroxyzine dihydrochloride1/2 | Midazolam&Hydroxyzine Dihydrochloride
Number analyzed (Participants) | 15 | 15 | 15
Number analyzed (number of orbital muscle/s, OCR occured) | 15 | 6 | 1
number of orbital muscle/s, OCR occured
  pausing surgery | 13 | 6 | 1
  atropin administration | 2 | 0 | 0
  cardiac resuscitation | 0 | 0 | 0

7. Other Pre Specified Outcome: The Orbital Muscle Name Which OCR Occurred During it's Traction
Description: The investigator records the orbital muscle name which OCR occurred during its traction; like Right eye medial rectus muscle, Right eye inferior oblique muscle, Right eye lateral rectus muscle, Left eye medial rectus muscle, Left eye inferior oblique muscle, Left eye lateral rectus muscle.
Time Frame: as for outcome 6
Population: The names of the orbital muscles which OCR occurred after traction was performed
Measure: Count of Units; unit: Orbital muscles which OCR occurred
Units Other Than Participants: Orbital muscles which OCR occurred
Arm/Group | Midazolam | Midazolam&Hydroxyzine dihydrochloride1/2 | Midazolam&Hydroxyzine Dihydrochloride
Number analyzed (Participants) | 15 | 15 | 15
Number analyzed (Orbital muscles which OCR occurred) | 15 | 6 | 1
Orbital muscles which OCR occurred
  Right eye medial rectus | 5 | 3 | 1
  Right eye lateral rectus | 3 | 0 | 0
  Left eye medial rectus | 6 | 2 | 0
  Left eye lateral rectus | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 day, during strabismus surgery(including anesthesia induction to emerge from anesthesia)
Description: regular investigator assessment
Groups:
- Midazolam: Demizolam, once on the operation day, usually ordered 15 minutes before strabismus operation by another anesthesiologist who is charged to perform anesthesia who is not related with the trial. The maximum dose of 0.5 mg/kg midazolam is given orally with cherry juice of maximum 5 ml. in Yeditepe University Hospital to the pediatric patients by the anesthesiologists.
  In all groups, patients are not selected to the groups and premedication and doses are not given by the investigator, they grouped according to the premedication given by the anesthesiologists, after the operation retrospectively.
  Midazolam: Demizolam 15mg/ml ampules, given orally with cherry juice
- Midazolam&Hydroxyzine Dihydrochloride: Midazolam and Hydroxyzine dihydrochloride, once on the operation day, usually ordered 15 minutes before strabismus operation by another anesthesiologist who is charged to perform anesthesia who is not related with the trial. The maximum dose of 0.5 mg/kg midazolam is given orally with the maximum dose of 1mg/kg hydroxyzine dihydrochloride in Yeditepe University Hospital to the pediatric patients by the anesthesiologists.
  In all groups patients are not selected to the groups and premedication doses are not given by the investigator, they grouped according to the premedication given by the anesthesiologists, after the operation retrospectively.
  Midazolam: Demizolam 15mg/ml ampules, given orally with cherry juice
  Hydroxyzine Dihydrochloride: Atarax 2mg/ml syrup, given orally
- Midazolam&Hydroxyzine dihydrochloride1/2: Midazolam and Hydroxyzine dihydrochloride, once on the operation day, usually ordered 15 minutes before strabismus operation by another anesthesiologist who is charged to perform anesthesia who is not related with the trial. The maximum dose of 0.5 mg/kg midazolam is given orally with hydroxyzine dihydrochloride (dose of 0.5 mg/kg) in Yeditepe University Hospital to the pediatric patients by the anesthesiologists.
  In all groups patients are not selected to the groups and premedication doses are not given by the investigator, they grouped according to the premedication given by the anesthesiologists, after the operation retrospectively.
  Midazolam: Demizolam 15mg/ml ampules, given orally with cherry juice
  Hydroxyzine Dihydrochloride: Atarax 2mg/ml syrup, given orally
Arm/Group | Midazolam | Midazolam&Hydroxyzine Dihydrochloride | Midazolam&Hydroxyzine dihydrochloride1/2
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
this current trial is not a prospective randomized study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03806270/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03806270/SAP_001.pdf